CLINICAL TRIAL: NCT02948816
Title: The Effects of Social Media on Food Intake and Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Prince Edward Island (Other)
Responsible Party: Principal Investigator, Travis Saunders, Assistant Professor, University of Prince Edward Island
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 6006850
Record Dates: First submitted 2016-10-24; First posted 2016-10-28 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Sedentary Lifestyle; Hunger; Eating
MeSH Terms: conditions — Sedentary Behavior | interventions — Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Facebook (Experimental): Participants will spend 30 minutes interacting with a Facebook page that is made up of 20% food-related posts, and 80% non food-related posts (news, sports, etc). They will be provided with bowls of snacks, which will be weighed before and after their session.
  Interventions: Behavioral: Facebook
- Facebook + Food (Experimental): Participants will spend 30 minutes interacting with a Facebook page that is made up of 70% food-related posts, and 30% non food-related posts (news, sports, etc). They will be provided with bowls of snacks, which will be weighed before and after their session.
  Interventions: Behavioral: Facebook + Food
- Colouring (Active Comparator): Participants will spend 30 minutes colouring. They will be provided with bowls of snacks, which will be weighed before and after their session.
  Interventions: Behavioral: Colouring

INTERVENTIONS:
Behavioral: Facebook — Participants will spend 30 minutes on a Facebook page that is primarily non-food related posts.
  Arms: Facebook
Behavioral: Facebook + Food — Participants will spend 30 minutes on a Facebook page that is food related posts.
  Arms: Facebook + Food
Behavioral: Colouring — Participants will spend 30 minutes colouring quietly.
  Arms: Colouring

SUMMARY:
Participants will be exposed to 3 conditions, in random order:

1. A Facebook page where 70% of posts are related to food.
2. A Facebook page where only 20% of posts are related to food.
3. A control condition (colouring quietly).

During each of the above conditions participants will be provided with identical snacks. The snacks will be weighed before and after each condition, to determine whether there is a change in food intake across the 3 conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25.

Exclusion Criteria:

* None

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10; Primary Completion 2017-04 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Ad libitum snack food intake | 30 minutes
  Participants will be provided with snack foods based on a previously completed food preference questionnaire. The food will be weighed before and after each session to determine caloric and macronutrient intake.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Prince Edward Island, Charlottetown, Prince Edward Island, Canada

IPD SHARING:
Plan to Share IPD: No